CLINICAL TRIAL: NCT06894459
Title: A Prospective, Multicenter, Multicohort Phase II Study: Evaluating the Efficacy and Safety of Preoperative Neoadjuvant Treatment With a PD-1 Inhibitor in Combination With Chemotherapy in Locally Advanced Laryngeal and Hypopharyngeal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRENT-003
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancers
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab; Cisplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- pCR group (Experimental): Patients with a pathological complete response (pCR) post-surgery receive adjuvant radiotherapy (50-56 Gy, 2.0 Gy/fraction).
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Nab-paclitaxel
- Non-pCR but without high-risk factors group (Experimental): Patients with non-pCR but without high-risk factors receive a combination of radiotherapy (56-60 Gy, 2.0 Gy/fraction) and cisplatin chemotherapy post-surgery.
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Nab-paclitaxel
- Non-pCR and high-risk factors group (Experimental): Patients with non-pCR and high-risk factors receive intensified radiotherapy (66-70 Gy, 2.0 Gy/fraction) along with cisplatin chemotherapy post-surgery.
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg, IV, 3 cycles
Drug: Cisplatin — cisplatin 75mg/m2, IV, 3 cycles
Drug: Nab-paclitaxel — Nab-paclitaxel 260mg, IV, 3 cycles

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) refers to a series of tumors that occur in the head and neck region, including the oral cavity, pharynx, larynx, nasal cavity, paranasal sinuses, thyroid gland, and salivary glands. Malignant tumors of the head and neck account for approximately 19.9% to 30.2% of all tumors in the body, ranking sixth in incidence among all malignant tumors, with over 90% being squamous cell carcinoma in terms of pathological type. The treatment of head and neck squamous cell carcinoma is primarily surgical. Early-stage cases can achieve a cure through simple surgical resection or radiotherapy. For locally advanced and late-stage cases, a combination of surgery with radiotherapy or chemotherapy can yield satisfactory therapeutic effects. However, most patients with head and neck tumors present at a locally advanced (Stage III to IVB) or late stage, possibly having lost the opportunity for surgery and can only opt for a comprehensive treatment mainly based on radiochemotherapy. Current data show that with standard treatment, the 5-year survival rates for patients with early-stage, locally advanced, and metastatic head and neck squamous cell carcinoma are 80%, 50%, and 25%, respectively. Fifty to sixty percent of newly diagnosed subjects cannot be cured and experience recurrence or metastasis within 3 years. For patients with recurrent or metastatic disease after first-line treatment failure, the median survival time with chemotherapy is only 6 to 9 months, with a 1-year survival rate of 5% to 33% and a 5-year survival rate of merely 3.6%. Laryngeal cancer and hypopharyngeal cancer hold unique significance among head and neck tumors because they not only threaten patients' lives but can also significantly affect their quality of life, particularly the preservation of laryngeal function. Laryngeal function includes voice production, swallowing, and breathing, and the loss of these functions can lead to a severe decline in quality of life. Traditionally, surgical resection has been the main treatment for these cancers, but total laryngectomy can result in permanent voice loss and significant psychological and social impacts. Therefore, how to effectively control the tumor while preserving laryngeal function has become an important goal of treatment.

PD-L1 is a key negative regulator of self-reactive T cells and plays a role in maintaining peripheral immune tolerance and suppressing autoimmunity in various ways, leading to T cell exhaustion and dysfunction, and allowing tumor cells to evade immune surveillance. PD-1/PD-L1 monoclonal antibodies restore the function of tumor-specific T cells by blocking the binding of PD-1 to PD-L1, thereby enhancing antitumor immunity and are now used to treat a variety of tumors. The efficacy of PD-1 inhibitors as neoadjuvant therapy in head and neck squamous cell carcinoma is not yet clear. However, given the good therapeutic effects of immunotherapy in head and neck squamous cell carcinoma, induction therapy with PD-1 inhibitors is considered to have promising clinical application prospects.

In summary, we hypothesize that compared with the traditional TPF (docetaxel, cisplatin, and fluorouracil) neoadjuvant chemotherapy regimen, a PD-1 inhibitor combined with chemotherapy regimen may be safer and more effective and easier to apply in clinical practice. At present, there are no reports of studies on the use of PD-1 inhibitors combined with chemotherapy regimens for locally advanced, resectable head and neck squamous cell carcinoma patients, either domestically or internationally. We plan to investigate the efficacy and safety of neoadjuvant treatment with PD-1 inhibitors combined with chemotherapy for resectable head and neck squamous cell carcinoma patients in China, to provide a basis for future neoadjuvant treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced laryngeal and hypopharyngeal squamous cell carcinoma who have been definitively diagnosed by histology and/or cytology, and whose TN staging meets: T1-4a, N0-3.
* No prior treatment received.
* Cisplatin-tolerant.
* Age ≥18 years.
* ECOG performance status of 0-1.
* Measurable disease as defined by RECIST v1.1.
* Normal organ function.
* Women and men of reproductive potential must agree to use appropriate contraceptive methods throughout the study period and for 180 days after the last study treatment.
* Male participants must not donate sperm during the entire study period and for 180 days after the last study treatment.

Exclusion Criteria:

* T stage is T4b.
* Presence of distant metastasis.
* Received live vaccines within 30 days prior to enrollment.
* Diagnosed with an immunodeficiency or received systemic corticosteroid treatment or any other form of immunosuppressive therapy within 7 days prior to enrollment.
* Have radiologically detectable (even if asymptomatic and/or previously treated) central nervous system metastases and/or carcinomatous meningitis.
* Have not fully recovered from surgery or from toxicities or complications due to interventions before starting the study.
* Have a history of allogeneic tissue/solid organ transplantation.
* Have had a severe hypersensitivity reaction (≥Grade 3) to PD-1 inhibitors, chemotherapy, or any of their excipients, or radiotherapy.
* Have an active autoimmune disease that has required systemic therapy within the past 2 years.
* Have a history of (non-infectious) pneumonitis that required treatment with corticosteroids.
* Have a history of infection with the Human Immunodeficiency Virus (HIV).
* Have a medical history that could confound study results or interfere with the participant during the study period.
* Have a known history of psychiatric disorders or substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival rate (2y-PFS rate) | 2 years
  To evaluate the 2y-PFS rate of neoadjuvant PD-1 inhibitors combined with chemotherapy in 3 arms; PFS was defined as the time from patient enrollment to the occurrence of the following events (local progression/recurrence or distant metastasis (including neoadjuvant stage) assessed by imaging or biopsy, death from any cause)

SECONDARY OUTCOMES:
Pathological complete response rate (pCR rate) | 3 months
  To evaluate the pCR rate of neoadjuvant PD-1 inhibitors combined with chemotherapy in 3 arms; pCR was defined as the absence of residual invasive squamous cell carcinoma cells in the resected primary tumor specimen and lymph nodes
Objective response rate (ORR) | 6 months
  To evaluate the ORR of neoadjuvant therapy with PD-1 inhibitors plus chemotherapy in 3 Arms; ORR is defined as The proportion of patients whose tumor volume shrinks to a pre-specified value and can be maintained for a certain period of time. It includes the proportion of patients with complete remission (CR) and partial remission (PR) to the total number of evaluable cases.
2-year overall survival rate (2y-OS rate) | 2 years
  To evaluate the 2y-OS rate of neoadjuvant PD-1 inhibitors plus chemotherapy in 3 Arms; OS was defined as the time from randomization until death from any cause.
Progression-Free Survival(PFS) | 2 years
  To evaluate the PFS of neoadjuvant PD-1 inhibitors plus chemotherapy in 3 arms in the overall population; PFS is defined as the length of time during and after treatment that a patient lives with a disease that does not get worse.
Incidence of Treatment-Emergent Adverse Events (TRAEs) of pembrolizumab combined with chemotherapy in neoadjuvant therapy | 3 years
  TRAEs include 5 levels, base on Common Terminology Criteria for Adverse Events (CTCAE) is widely accepted as the standard classification and severity grading scale for adverse events in cancer therapy, clinical trials and other oncology settings.

IPD SHARING:
Plan to Share IPD: No